CLINICAL TRIAL: NCT05653089
Title: Evaluation of Actions to Improve Positioning in Wheelchaire Bound Patients at Risk of Slipping : Pilot Study
Brief Title: Positioning in Wheelchair Bound Patients
Acronym: AAPO'G
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: FondationbHopale (Other)
Collaborators: GHICL (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HOP-RIPH2-21-05
Record Dates: First submitted 2022-11-10; First posted 2022-12-16 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-04

CONDITIONS: Neurological Disease
Keywords: wheelchair; seating discomfort
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients meeting the study eligibility criteria (Experimental)
  Interventions: Procedure: Choice and adjustment of the wheelchair according to the patient's needs

INTERVENTIONS:
Procedure: Choice and adjustment of the wheelchair according to the patient's needs — After a personalized analysis of the patient and his needs, the occupational therapists define the equipment necessary for the good positioning of the patient:
  * Choice and adjustments of the wheelchair
  * Choice and adjustments of the wheelchair/patient interface

SUMMARY:
The choice of the most suitable chair as well as the improvement of the patient's positioning on this wheelchair is important to limit the discomfort, to prevent the risks of bedsores, the pains related to prolonged sitting and finally to support the interaction of the patient with its environment. The goal of this prospective, longitudinale, monocentric study is to evaluate the impact of standardized positioning in wheelchair-bound patients at risk of slipping.

The main questions on the positioning actions are:

* their actions impact of positioning actions on shear forces
* their impact on sliding in the chair
* their impact on the feeling of discomfort in the chair
* their impact on the caregivers' feelings about the patient's difficulties (eating, transfers, sliding)

Participation in this study will involve an increase in the number of transfers required for shear sheet placement and removal, as well as the time required for ischial measurement and the time to complete the (Tool for Assessing Wheelchair disComfort) TAWC questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized for a minimum of 9 days (minimum 48-hour reflection period after information)
* Patient aged between 18 and 80 years,
* Patient with a sitting time in a wheelchair > or equal to 1 hour,
* Patient with a neurological condition : multiple sclerosis, stroke, spinal cord injury, Parkinson disease, neurodegenerative diseases...
* Patient informed of the study and having given his written consent,

Non inclusion Criteria:

* Cognitive disorders that do not allow the understanding of instructions
* Patient with a pressure sore
* Pregnant or breastfeeding woman
* Patient under legal protection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-22 (Estimated)

PRIMARY OUTCOMES:
Evolution of shear measurement with the Shear® sensor | Day 0 therefore before the implementation of the positioning actions then at Day 1 and Day 7
  Shear will be measured over a period of one hour (shear evolution over one hour), during which the patient will follow a standardized activity program.

SECONDARY OUTCOMES:
Comparison of the sliding distance | Day 0 therefore before the implementation of the positioning actions then at Day 1 and Day 7
  The sliding distance is measured by the position of the ischiums. It is the difference between the position measured before and after 1 hour of standardized activities.
Evolution of the score on the TAWC scale | Day 0 therefore before the implementation of the positioning actions then at Day 7
  The TAWC (Tool for Assessing Wheelchair discomfort) scale assesses 2 discomfort scores:
  * an assessment of general discomfort, based on 13 items scored on 7 points
  * an evaluation of the intensity of the discomfort, based on 9 items from 0 to 10.
Evolution of the caregiver questionnaire score (Likert scale) | Day 0 therefore before the implementation of the positioning actions then at Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Jean Gabriel PREVINAIRE, MD, Principal Investigator — Fondation Hopale
Locations (1):
- Julien PAGER, Berck, Hauts-de-France, France

IPD SHARING:
Plan to Share IPD: No